CLINICAL TRIAL: NCT06310343
Title: A Study of a New Assay to Detect Anti-drug Antibodies to Alemtuzumab and Their Potential Impact in Multiple Sclerosis
Brief Title: ADAs to Alemtuzumab
Status: Active, not recruiting | Type: Observational
Sponsor: Queen Mary University of London (Other)
Responsible Party: Sponsor
Other Study IDs: 304993
Record Dates: First submitted 2024-03-07; First posted 2024-03-15 (Actual); Last update posted 2025-03-17 (Actual); Status verified 2025-03

CONDITIONS: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis | interventions — Alemtuzumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Alemtuzumab — Licensed dose

SUMMARY:
The main aim is to quantify the changes in alemtuzumab antibody-anti-alemtuzumab over a 24 months period

DETAILED DESCRIPTION:
Primary To quantify the longitudinal changes in alemtuzumab ADAs over a 24 month period.

Secondary

1. Relative occurrence of infusion-related reactions based on high alemtuzumab ADA levels prior to course 2.
2. Relative change in lymphocyte counts after the second infusion of alemtuzumab in ADA positive patients to assess the health economic impact of infusion-related reactions.
3. Relative change in relapses or EDSS score based on alemtuzumab ADA levels to assess the health economic impact of disease activity.
4. Relative change in relapses or EDSS score based on alemtuzumab ADA levels.
5. Relative change in T2 lesion number or Gd-enhancing lesions, and serum NfL based on alemtuzumab ADA levels to assess the health economic impact of disease activity.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with RRMS who are being treated with alemtuzumab at Barts Health NHS Trust will be approached to participate in the study.
2. Patients must be willing and able to undergo blood tests.

Exclusion Criteria:

1. Ineligible for alemtuzumab under NHS England prescribing guidelines.
2. Those unable to comply with study requirements, including frequency of visits. Abnormal baseline investigations (WBC<3 x 10*9/l, lymphocytes <1.0 x 10*9/l, neutrophil count <1.5 x 10*9/l, platelet count <100 x 10*9/l, haemoglobin <110 g/l, LFT >/3x upper limit of normal of site reference ranges, potassium <2.8 mmol/l or >5.5 mmol/l, sodium /,125 mmol/l, creatinine >130 umol/l).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Relapsing-remitting MS
Sampling Method: Non-Probability Sample
Enrollment: 15 (Actual)
Dates: Start 2022-07-12 (Actual); Primary Completion 2025-11-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
To quantify the longitudinal changes in alemtuzumab ADAs | 2 years

SECONDARY OUTCOMES:
1. Relative occurrence of infusion-related reactions based on high alemtuzumab ADA levels prior to course 2. | 1 year
2. Relative change in lymphocyte counts after the second infusion of alemtuzumab in ADA positive patients to assess the health economic impact of infusion-related reactions. | 2 years
3. Relative change in relapses or EDSS score based on alemtuzumab ADA levels to assess the health economic impact of disease activity. | 2 years
4. Relative change in relapses or EDSS score based on alemtuzumab ADA levels | 2 years
5. Relative change in T2 lesion number or Gd-enhancing lesions, and serum NfL based on alemtuzumab ADA levels to assess the health economic impact of disease activity. | 2 years

CONTACTS AND LOCATIONS:
Locations (1):
- Barts Health NHS Trust, London, Second Floor Neurophys Dept, United Kingdom

IPD SHARING:
Plan to Share IPD: No